CLINICAL TRIAL: NCT06792058
Title: Comparative Study of TetraGraph and Mechanomiograph Neuromuscular Monitors in Clinical Settings
Acronym: EMGvsMMG
Status: Completed | Type: Observational
Sponsor: University of Debrecen (Other)
Responsible Party: Principal Investigator, Tamas Vegh, MD, MD PhD, University of Debrecen
Other Study IDs: AITT 2023/10
Record Dates: First submitted 2025-01-14; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Patients Undergoing General Anesthesia
Keywords: Neuromuscular monitoring; MMG; EMG

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- 20 surgical patients: 20 patients undergoing surgical procedures and receiving muscle relaxation
  Interventions: Device: Mechanomiograph: The "gold standard" of quantitative monitoring; Device: Electromiograph

INTERVENTIONS:
Device: Mechanomiograph: The "gold standard" of quantitative monitoring — The "gold standard" of quantitative monitoring is mechanomyography (MMG), which measures the force of contraction of the adductor pollicis muscle following ulnar nerve stimulation. MMG responses are accurate and reproducible. However, the complex and bulky devices are only suitable for research use, are not suitable for clinical use and are not commercially available.
Device: Electromiograph — Another type of monitor is the electromyograph, which can be seen as an alternative to mechanomyography because of its accuracy. This technique measures muscle activity as a summation of the action potentials of muscle fibres. This activity is proportional to the strength of the muscle contraction. The most commonly innervated nerve is also the ulnar nerve, which innervates the abductor digiti minimi and the first dorsalis interosseus muscles. During the measurements, electrical signals from these muscles are detected. EMG has several advantages over other monitoring techniques. It does not require immobilisation of the hand, thumb immobility is not a problem, no preload is required, and hypothermia does not affect the hand as much as other neuromuscular monitors. The TetraGraph (Senzime AB, Sweden) is a portable EMG-based neuromuscular minitor for which the manufacturers received marketing approval from the U.S. Food and Drug Administration (FDA) in 2019.

SUMMARY:
Background: Neuromuscular monitoring plays a critical role in reducing postoperative residual neuromuscular blockade (PRNB), a significant risk factor for respiratory complications. Despite the availability of various monitoring techniques, the validation of newer devices remains an ongoing challenge. This study compares the performance of the electromyography (EMG)-based Tetragraph neuromuscular monitor with the gold standard mechanomyography (MMG) device, focusing on their accuracy and reliability in clinical settings.

Methods: Twenty cases were conducted during general surgeries requiring neuromuscular relaxation. Ulnar nerve was stimulated via the Tetragraph which detected the compound muscle action potential (CMAP) of adductor pollicis muscle. Simultaneously on the same arm the isometric force of the same stimulated muscle was registrated by the MMG and displayed in the Labchart 8 program. Bland-Altman analysis was used to describe the agreement between devices during distinct phases of neuromuscular blockade. The primary endpoint of the study was the comparison of TOF values of MMG and EMG during induction. In recovery, two groups were made from TOFRs: below and above the recommended muscle recovery to exclude PRNB (TOFR≥90%) (Fuchs-Buder 2023). Additionally, in deeper neuromuscular blockade Train-of-Four Count (TOFC), and Post-Tetanic Count (PTC) values were also analysed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over.
* ASA (American Society of Anesthesiology) physical status I-III.
* Informed written consent.
* Surgery requires the use of a moderate-duration muscle relaxant.

Exclusion Criteria:

* History of neuromuscular disease (e.g. stroke with hemi symptoms, myasthenia gravis, severe polyneuropathy).
* Medication affecting neuromuscular transmission.
* Open wound or rash due to electrode position
* Expected difficult intubation.
* Pregnancy, breast-feeding.
* Implanted pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing general surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
concordance of the two devices | Intraoperativ
  The primary endpoint of the study is the comparison of TOF values measured by mechanomyography and electromyography, and the examination of the measurement concordance of the two devices.

CONTACTS AND LOCATIONS:
Overall Officials: László Asztalos, PhD, Study Director — University of Debrecen, Faculty of Medicine, Department of Anaesthesiology and Intensive Care
Locations (1):
- University of Debrecen, Department of Anesthesiology and Intensive Care, Debrecen, Hajdú-Bihar, Hungary

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fuchs-Buder T, Claudius C, Skovgaard LT, Eriksson LI, Mirakhur RK, Viby-Mogensen J; 8th International Neuromuscular Meeting. Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision. Acta Anaesthesiol Scand. 2007 Aug;51(7):789-808. doi: 10.1111/j.1399-6576.2007.01352.x. PMID 17635389
- [Background] Sato H, Iwasaki H, Doshu-Kajiura A, Katagiri S, Takagi S, Luthe SK, Suzuki T. Comparison of two electromyography-based neuromuscular monitors, AF-201P and TetraGraph, in rocuronium-induced neuromuscular block: A prospective comparative study. Anaesth Crit Care Pain Med. 2022 Dec;41(6):101145. doi: 10.1016/j.accpm.2022.101145. Epub 2022 Aug 31. PMID 36057386
- [Background] Nemes R, Lengyel S, Nagy G, Hampton DR, Gray M, Renew JR, Tassonyi E, Fulesdi B, Brull SJ. Ipsilateral and Simultaneous Comparison of Responses from Acceleromyography- and Electromyography-based Neuromuscular Monitors. Anesthesiology. 2021 Oct 1;135(4):597-611. doi: 10.1097/ALN.0000000000003896. PMID 34329371
- [Background] Kopman AF, Justo MD, Mallhi MU, Abara CE, Neuman GG. The influence of changes in hand temperature on the indirectly evoked electromyogram of the first dorsal interosseous muscle. Can J Anaesth. 1995 Dec;42(12):1090-5. doi: 10.1007/BF03015094. PMID 8595683
- [Background] Engbaek J, Skovgaard LT, Friis B, Kann T, Viby-Mogensen J. Monitoring of the neuromuscular transmission by electromyography (I). Stability and temperature dependence of evoked EMG response compared to mechanical twitch recordings in the cat. Acta Anaesthesiol Scand. 1992 Aug;36(6):495-504. doi: 10.1111/j.1399-6576.1992.tb03506.x. PMID 1325093
- [Background] Naguib M, Brull SJ, Johnson KB. Conceptual and technical insights into the basis of neuromuscular monitoring. Anaesthesia. 2017 Jan;72 Suppl 1:16-37. doi: 10.1111/anae.13738. PMID 28044330
- [Background] Naguib M, Kopman AF, Ensor JE. Neuromuscular monitoring and postoperative residual curarisation: a meta-analysis. Br J Anaesth. 2007 Mar;98(3):302-16. doi: 10.1093/bja/ael386. PMID 17307778
- [Background] Todd MM, Hindman BJ, King BJ. The implementation of quantitative electromyographic neuromuscular monitoring in an academic anesthesia department. Anesth Analg. 2014 Aug;119(2):323-331. doi: 10.1213/ANE.0000000000000261. PMID 24878683
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS. Residual neuromuscular blockade and critical respiratory events in the postanesthesia care unit. Anesth Analg. 2008 Jul;107(1):130-7. doi: 10.1213/ane.0b013e31816d1268. PMID 18635478
- [Background] Berg H, Roed J, Viby-Mogensen J, Mortensen CR, Engbaek J, Skovgaard LT, Krintel JJ. Residual neuromuscular block is a risk factor for postoperative pulmonary complications. A prospective, randomised, and blinded study of postoperative pulmonary complications after atracurium, vecuronium and pancuronium. Acta Anaesthesiol Scand. 1997 Oct;41(9):1095-1103. doi: 10.1111/j.1399-6576.1997.tb04851.x. PMID 9366929
- [Background] Arbous MS, Meursing AE, van Kleef JW, de Lange JJ, Spoormans HH, Touw P, Werner FM, Grobbee DE. Impact of anesthesia management characteristics on severe morbidity and mortality. Anesthesiology. 2005 Feb;102(2):257-68; quiz 491-2. doi: 10.1097/00000542-200502000-00005. PMID 15681938
- [Background] Eriksson LI. Reduced hypoxic chemosensitivity in partially paralysed man. A new property of muscle relaxants? Acta Anaesthesiol Scand. 1996 May;40(5):520-3. doi: 10.1111/j.1399-6576.1996.tb04482.x. PMID 8792879
- [Background] Sundman E, Witt H, Olsson R, Ekberg O, Kuylenstierna R, Eriksson LI. The incidence and mechanisms of pharyngeal and upper esophageal dysfunction in partially paralyzed humans: pharyngeal videoradiography and simultaneous manometry after atracurium. Anesthesiology. 2000 Apr;92(4):977-84. doi: 10.1097/00000542-200004000-00014. PMID 10754616
- [Background] Eriksson LI, Sato M, Severinghaus JW. Effect of a vecuronium-induced partial neuromuscular block on hypoxic ventilatory response. Anesthesiology. 1993 Apr;78(4):693-9. doi: 10.1097/00000542-199304000-00012. PMID 8096684
- See also: The tetragraph manufacturer's website. — https://www.senzime.com/en/tetragraph